CLINICAL TRIAL: NCT06055049
Title: The Effect of Kinesio Taping on Pain, Stress, Sleep and Quality of Life in University Students With Primary Dysmenorrhea: A Randomized Controlled Study
Brief Title: Effects of Kinesio Tape in Primary Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yağmur SÜRMELİ (Other)
Responsible Party: Sponsor-Investigator, Yağmur SÜRMELİ, Lecturer, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-41901325-200-57905 2023/016
Record Dates: First submitted 2023-09-18; First posted 2023-09-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea Primary; Kinesio Taping; Pain; Stress; Sleep Quality; Quality of life
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders | interventions — Methods; Population Groups

STUDY DESIGN:
Intervention Model Description: There will be 2 groups (kinesio taping and sham taping) and each group will consist of at least 28 people.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping (n=28) (Experimental): Kinesio taping certified researcher Y.S. It will be implemented by. Kinesio Taping will be applied to the study group participants during three menstrual cycles. Kinesio taping will be done face to face by the researcher in the laboratory. The participants were given the "Mcgill Pain Scale Short Form", "Menstruation Symptom Scale", "Perceived Stress Scale", "Pittsburgh Sleep Quality Index" and "World Health Organization Quality of Life Scale-Short Form (WHOQOL-BREF-TR) " immediately after the third cycle and the fourth cycle without treatment. will be applied. The follow-up of the implementation process will be recorded with the MSF and KBIF prepared by the researcher.
  Kinesio tapes will be applied to the sacral area with 100% tension twice a week, starting from the first start of menstruation. It will continue like this until the end of the 3rd period of menstruation.
  Interventions: Other: Intervention (Kinesio Taping) group
- Sham Taping (n=28) (Placebo Comparator): Sham taping (fake or tensionless kinesio taping) will be applied to students in the placebo group. The quality of the kinesio tape used in sham taping will be the same. "Mcgill Pain Scale Short Form", "Menstruation Symptom Scale", "Perceived Stress Scale", "Pittsburgh Sleep Quality Index" and "World Health Organization Quality of Life Scale-Short Form (WHOQOL-BREF-TR) administered to participants in the placebo group before the first session )" will be refilled at the end of the third cycle and at the end of the fourth cycle without treatment. In order to eliminate the ethical problems that may occur in the control group, kinesio taping will be applied to the participants in this group after the data collection process of the research is completed.
  Kinesio tapes will be applied to the sacral area without tension, twice a week, starting from the first start of menstruation. This situation will continue until the end of the 3rd menstrual period.
  Interventions: Other: Intervention (Kinesio Taping) group

INTERVENTIONS:
Other: Intervention (Kinesio Taping) group — It is the group to which Kinesio Taping applied.

SUMMARY:
The purpose of this [study type: a single-blind, placebo-controlled randomization study] was to determine the effect of kinesio taping on pain, stress, sleep, and quality of life in college students with primary dysmenorrhea. The key question(s) it aims to answer are:

• [Is there a difference between pain, stress, sleep quality and quality of life scores in the post-kinesio taping intervention group and the placebo group?] Participants [both groups will come to the laboratory to replace their kinesio bands on the specified dates] If there is a comparison group: Researchers will compare with the placebo group.

DETAILED DESCRIPTION:
The opinion of a biostatistician was taken to determine the population of volunteers in the study. As a result of this opinion, 1st year female students who enroll in Toros University Vocational School of Health Services in the 2023-2024 Fall Semester will form the universe of the research. The sample of the study consisted of 56 volunteers who were 18 years of age and older, who met the inclusion criteria, had a Visual Analog Scale (VAS) score of four and above, a Menstruation Symptom Scale score of 60 and above, and had primary dysmenorrhea (Kinesio tape applied: 28 students, sham The band applied: 28 students will be formed After the female students to be included in the sample are determined, their assignments to the study and control groups will be made according to the randomization method. The research will start in the fall semester of the 2023-2024 academic year and the data collection period is planned as 4 months (25.09.2023-25.01.2024).

Before starting the application to the students in the study group, the researcher Y.S. Fast and easy application steps will be explained with the demonstration method, supported by visual presentations.

Kinesio Taping will be applied to the study group participants during three menstrual cycles. Kinesio taping will be done face to face by the researcher in the laboratory. The participants were given the "Mcgill Pain Scale Short Form", "Menstruation Symptom Scale", "Perceived Stress Scale", "Pittsburgh Sleep Quality Index" and "World Health Organization Quality of Life Scale-Short Form" immediately after the third cycle and the fourth cycle without treatment. -BREF-TR)" will be applied. The follow-up of the implementation process will be recorded with the MSF and KBIF prepared by the researcher.

Sham taping (fake or tensionless kinesio taping) will be applied to students in the placebo group. The quality of the kinesio tape used in sham taping will be the same. "Mcgill Pain Scale Short Form", "Menstruation Symptom Scale", "Perceived Stress Scale", "Pittsburgh Sleep Quality Index" and "World Health Organization Quality of Life Scale-Short Form (WHOQOL-BREF-TR) administered to participants in the placebo group before the first session )" will be refilled at the end of the third cycle and at the end of the fourth cycle without treatment. In order to eliminate the ethical problems that may occur in the control group, kinesio taping will be applied to the participants in this group after the data collection process of the research is completed.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old,
* 1st grade student
* Willing to participate in the research,
* Open to communication,
* Having a regular menstrual period (occurring at intervals of 21-35 days and lasting 3-8 days),
* Menstrual pain severity is at least 4 according to the Visual Pain Scale,
* A score of 60 or more on the Menstruation Symptom Scale,
* Not using hormonal contraception and intrauterine device,
* Not pregnant and not experiencing pregnancy before,
* Does not have a systemic and chronic disease,
* Have not had a gynecological disorder or surgical operation before,
* Not using analgesics 6 hours before and during the study period,
* Not regularly applying kinesio taping,
* Students without psychiatric problems.

Exclusion Criteria:

* under the age of 18,
* Studying in the 2nd grade,
* Not willing to participate in the research,
* Closed to communication,
* Not having a regular menstrual period (not occurring at intervals of 21-35 days and lasting more or less than 3-8 days),
* Menstrual pain severity is less than 4 according to the Visual Pain Scale,
* A score below 60 on the Menstruation Symptom Scale,
* Using hormonal contraception and intrauterine device,
* who are pregnant and have experienced pregnancy before,
* Having a systemic and chronic disease,
* Having had a gynecological disorder or surgical operation before,
* Using analgesics 6 hours before and during the study period,
* Regularly applying kinesio taping, Students with psychiatric problems.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The female just have dysmenhorea
Enrollment: 56 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Mcgill Pain Scale | Before the study (Pre-test) 2. End of the application (week 12) 3. Post-test (at the end of the 16. week).
  Mcgill Pain Scale Short Form (MAS-SF) The Mcgill Pain Scale Short Form was developed by Ronald Melzack in 1987 to determine the nature, effect, and overall pain intensity of pain.
  In the first part of the Mcgill Pain Scale Short Form, there are 15 word groups describing the sensory/perceptual pain dimension (first 11 words) and emotional/emotional pain dimension (last four words).
  In the second part of the scale, the severity of the pain at that moment is determined from the patient by using the VAS.
  In the third part of the scale, a six-point Likert type scale is used to determine the general pain intensity. Scale; It consists of expressive values ranging from 0 = no pain, 1 = mild, 2 = bothersome, 3 = distressing, 4 = terrible, 5 = unbearable pain.
VAS pain scale | Pre-Study will be applied to determine compliance with the criteria.
  Visual Analogue Scale (VAS)
  Different scales are used in studies to measure the level of pain. In our study, the pain intensity of the participants will be determined by using the Visual Analogue Scale (VAS) in the Determination of Compliance with the Criteria Form. VAS has been developed in order to be able to specify the severity of pain more easily by converting some values that cannot be measured numerically. VAS is a safe, easily applicable measurement tool that has been generally accepted in the world literature for many years. A low score on the VAS indicates low/low pain intensity, and a high score indicates high/severe pain.
Menstrual Symptom Questionnaire | Before the study (Pre-test) 2. End of the application (week 12) 3. Post-test (at the end of the 16. week).
  Menstrual Symptom Questionnaire (MSQ) Menstruation Symptom Scale (MSI) It was developed by Chesney and Tasto in 1975 to assess menstrual pain and symptoms . The scale, which is a five-point Likert type and consists of 24 items, was updated by Negriff et al. in 2009 by re-evaluating its factor structure and usability. The MSÖ score is calculated by taking the total mean score of the items in the scale. An increase in the mean score indicates an increase in the severity of menstrual symptoms. The score obtained from the sub-dimensions in the scale is calculated by taking the total score average of the items in the sub-dimensions. An increase in the mean score for the sub-dimensions indicates an increase in the severity of menstrual symptoms related to that sub-dimension.
Adaptation of the Perceived Stress Scale | Before the study (Pre-test) 2. End of the application (week 12) 3. Post-test (at the end of the 16. week).
  Adaptation of the Perceived Stress Scale (Pss-14) The Perceived Stress Level Scale was focused on by Cohen, Kamarck, and Mermelstein in 1983 to determine perceived stress controls. The Turkish validity and reliability study of the scale was conducted by Eskin et al. This 14-item scale reflects the extent to which people perceive purposive stress according to the basic idea in their lives. The scale is 5-point Likert type (0: Never, 1: Almost Never, 2: Sometimes, 3: Often, 4: Very Often). is a scale. One of the questions in the scale is to evaluate the changes in mood in the last month. There are seven items (4, 5, 6, 7, 9, 10 and 13) containing positive statements in the scale and these items are scored in reverse. The stress level perceived by the respondent is determined by adding the scores obtained from the items. A score between 0-56 points is taken in the scale. The higher the score, the higher the perceived stress level. The Cronbach Alpha Coefficient of the scale is 0.84.
Pittsburgh Sleep Quality Index | Before the study (Pre-test) 2. End of the application (week 12) 3. Post-test (at the end of the 16. week).
  Pittsburgh Sleep Quality Index (PUKI) PSQI assesses sleep quality over the past month. 19 out of 24 questions in PSQI are self-report questions. Five questions are answered by the spouse or roommate. The last five questions are for clinical information purposes only and are not included in the scoring. Self-report questions involve several factors related to sleep quality. These relate to the estimation of sleep duration, sleep latency, and the frequency and severity of certain sleep-related problems. Subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction were divided into 18 items included in the scoring. Each item is evaluated over 0-3 points. As the total score obtained from the scale increases, sleep quality decreases. Patients with a total score of 0-4 on PUKI are classified as having good sleep quality. Scale scores of 5 and above indicate poor sleep quality.
World Health Organization Quality of Life Scale Short Form | Before the study (Pre-test) 2. End of the application (week 12) 3. Post-test (at the end of the 16. week).
  World Health Organization Quality of Life Scale (WHOQOL-BREF-TR) The World Health Organization Quality of Life Scale-Short Form was developed by the World Health Organization (WHO) in 1998 to assess the quality of life of individuals. The Turkish validity and reliability studies of the scale were carried out by Eser et al. WHOQOL-BREF-TR consists of 27 questions and item 27 is not usually included in statistical analysis. The scale does not have a total score, each dimension is evaluated within itself. The scores of the dimensions are evaluated between 4-20. Increasing score indicates goodness.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu VEFIKULUCAY YILMAZ, Prof, Study Chair — Mersin University Faculty of Nursing; Yagmur SURMELI, Lect., Principal Investigator — Mersin University Faculty of Nursing
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No